CLINICAL TRIAL: NCT00732602
Title: The Effects of GIP and GLP-2 on the Secretion of Glucagon in Patients With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Mikkel Christensen MD, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: H-D-2007-0058
Record Dates: First submitted 2008-08-11; First posted 2008-08-12 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Diabetes Mellitus
Keywords: Glucagon; Glucose-dependent Insulinotropic Polypeptide; Glucagon-Like peptide 2
MeSH Terms: conditions — Diabetes Mellitus | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- B (Active Comparator): GLP-2 infusion
  Interventions: Other: GLP-2 infusion
- C (Placebo Comparator): Sodium-chloride infusion
  Interventions: Other: Sodium-chloride
- A (Active Comparator): GIP-infusion
  Interventions: Other: GIP-infusion

INTERVENTIONS:
Other: GIP-infusion
  Arms: A
Other: Sodium-chloride
  Arms: C
Other: GLP-2 infusion
  Arms: B

SUMMARY:
The purpose of this study is to determine whether Glucose-dependent Insulinotropic Polypeptide (GIP) or Glucagon Like Peptide 2 (GLP-2) has an affect on the secretion of Glucagon from the pancreas in patients with type 1 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Caucasians over 18 years with type 1 diabetes (WHO criteria)
* Arginine test without rise in plasma C-peptide
* Normal blood Hemoglobin
* Informed consent

Exclusion Criteria:

* Liver disease
* Diabetic nephropathy
* Treatment with medications unpausable for 12 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-01; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
plasma-glucagon Area Under Curve at 0-90 min. and 90-180 min.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Gentofte, Hellerup, Capital Region, Denmark